CLINICAL TRIAL: NCT06026501
Title: A Phase Ib/II Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of PE0116 and PE0105 Injection in Treatment of Patients With Advanced Solid Tumor
Brief Title: A Phase Ib/II Clinical Trial of PE0116 and PE0105 Injection in Treatment of Patients With Advanced Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Collaborators: Shanghai HyaMab Biotech Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-0116-002
Record Dates: First submitted 2023-08-15; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PE0116+PE0105 (Experimental): PE0116 injection will be given 1mg/kg or 2mg/kg every three weeks and PE0105 injection will be given 3mg/kg every threee weeks until there appears evidence of progressive disease, intolerable toxicity, or the patient discontinues from the study treatment for other reasons.
  Interventions: Drug: PE0116,PE0105

INTERVENTIONS:
Drug: PE0116,PE0105 — 1. PE0116: 4-1BB Agonist Antibody Drug
  2. PE0105: PD-1 Monoclonal Antibody Drug
  Other Names: PE0116 injection，PE0105 injection

SUMMARY:
This study is a one-arm, open, multicenter phase 1b/2 clinical trial of PE0116combined with PE0105 in patients with Advanced Solid Tumors, aiming at exploring the MTD and RP2D and observing the preliminary efficacy.The trial can be divided into two parts: dose escalation part and expansion part.PE0105 is administered as a fixed-dose intravenous injection(3mg/kg Q3w）.

DETAILED DESCRIPTION:
Phase Ib

This is a dose escalation,3+3 design study, to evaluate the safety and tolerability, and to determine the RP2D of PE0116 injection in patients with advanced solid tumors. One cycle is 21 days.

Phase II

This is an expansion phase in patients with advanced solid tumors such as ovarian cancer, cervical cancer, renal cancer, head and neck cancer to further evaluate the safety, tolerability and preliminary anti-tumor activity of PE0116 injection at the RP2D combined with PE0105 injection every three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily sign the informed consent form, understand the study and are willing to follow and able to complete all study procedures,
2. Male or female, 75 ≥ age ≥ 18 years,
3. Patients enrolled in Phase Ib are those with histopathologically or cytologically confirmed metastatic or unresectable locally advanced, recurrent solid tumors (ovarian cancer, cervical cancer, renal cancer, head and neck cancer, etc.) who have failed to respond to or are intolerant to standard treatment regimens or have no standard effective treatment regimen, and at least one evaluable lesion meeting the definition of RECISTv1.1,
4. Patients enrolled in Phase II must have at least 1 measurable lesion consistent with the definition of RECISTv1.1 and need to meet one of the following tumor types: a).histologically and/or cytologically confirmed diagnosis of advanced renal cancer, head and neck cancer, or cervical cancer who have failed at least 1 line of prior therapy with PD-1 and anti-PD-1/PD-L1 antibodies alone or in combination with chemotherapy; failure of anti-PD-1/PD-L1 antibodies is defined as disease progression after achieving complete response (CR) or partial response (PR) with anti-PD-1/PD-L1 antibodies alone or in combination with chemotherapy, or disease progression after ≥ 6 months of stable disease (SD); b). histologically and/or cytologically confirmed diagnosis of ovarian cancer who have received 1 line of prior therapy consisting of at least 1 platinum agent and imaging evidence of disease progression within 6 months of the last dose of platinum-based chemotherapy,
5. Patients who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1,
6. Patients who have a life expectancy of at least 3 months,
7. Patients who are ≥ 4 weeks after receiving anti-tumor therapy, such as chemotherapy, radiotherapy, biotherapy, endocrine therapy and immunotherapy before the first dose of study drug,
8. Patients need to have appropriate organ and hematopoietic function, laboratory tests，
9. Male and female patients of childbearing potential should agree to use effective contraception from the signing of the informed consent form until 3 months after the last dose.

Exclusion Criteria:

1. Patients with clinically symptomatic central nervous system metastases and/or carcinomatous meningitis,
2. Patients who have previously failed to recover from adverse reactions to CTCAE V5.0 grade ≤ 1,
3. Uncontrolled stable systemic disease with treatment，
4. Any active autoimmune disease or documented autoimmune disease, or systemic syndrome previously requiring systemic steroids or immunosuppressive drugs，
5. Patients who require systemic corticosteroids (at doses equivalent to > 10 mg prednisone/day) or other immunosuppressive drugs within 14 days before enrollment or during the study，
6. History of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation, or stem cell transplantation，
7. Patients who have pulmonary tuberculosis and are in active phase at screening，
8. Patients with active chronic hepatitis B or active hepatitis C，
9. Patients who have received anti-4-1BB target drugs，
10. Known subjects who have previously treated with macromolecular protein agents/monoclonal antibodies, or known to have a serious allergic reaction to any component of the test drug (CTCAE V5.0 grade greater than 3)，
11. Patient plan to have major surgery during this study including a 28-day screening period，
12. Severe infection within 4 weeks before the first dose,Or patients with active infection requiring intravenous antibiotics within the first 2 weeks,
13. Patient participated in other clinical trials of drugs within 4 weeks before enrollment and have been enrolled in drug therapy, or did not reach 4 weeks after the end of treatment (EOT),
14. Patient had a history of alcoholism, drug abuse or drug abuse within the past 1 year,
15. Patien had ≥ grade 3 irAEs or ≥ grade 2 immune-related myocarditis in previous immunotherapy,
16. Patient had a history of other primary malignancies ,
17. Patient had a history of moderate or severe dyspnea at rest due to advanced malignancies or their complications or severe primary lung disease, or currently required continuous oxygen therapy, or currently had interstitial lung disease (ILD) or pneumonia,
18. Patient received live attenuated vaccines within 4 weeks before the first dose or planned to receive during the study,
19. Patient had a clear history of neurological or psychiatric disorders, such as epilepsy, dementia, and poor compliance,
20. Patient was pregnant or lactating women; Eligible patients of childbearing potential (men and women) did not agree to use a reliable method of contraception during the trial and for at least 3 months after the last dose, and female patients of childbearing age had a positive blood or urine pregnancy test within 7 days before enrollment,
21. Patients who were considered by the investigator to be unsuitable for participation in the trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated by NCI-CTCAE v5.0 | From time of first dose to 21 days after the first dose.
  Incidence of dose limited toxicities and associated dose of PE0105 and PE0116
Adverse events evaluated by NCI CTCAE v5.0 | From time of first dose to 90 days after the last dose.
  Incidence of adverse events and associated dose of PE0105 and PE0116
Recommended Phase 2 Dose | From time of first dose of the first patient to the last dose of the last patient in phase 1b..
  Recommended dose for phase II clinical trial is explored through dose escalation in phase Ib clinical trial.
Objective response rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  The proportion of subjects who have a Complete Response or Partial Response

SECONDARY OUTCOMES:
Disease control rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  The proportion of subjects who have a Complete Response or Partial Response
Plasma concentration of PE0116 and PE0105 | From one hour before the first dose to 90 days after the last dose.
  This composite endpoint will measure the plasma concentration of PE0116 and PE0105.